CLINICAL TRIAL: NCT01743248
Title: Evaluation of the Influence of Psychological Factors on Balance Control Compensation After Vestibular Schwannoma Surgery
Brief Title: Vestibular Schwannoma and Psychological Factors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: University of Lorraine (Other)
Responsible Party: Principal Investigator, Cecile PARIETTI-WINKLER, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2012-A00522-41
Record Dates: First submitted 2012-09-28; First posted 2012-12-06 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Vestibular Schwannoma
Keywords: vestibular schwannoma; balance; psychological factors
MeSH Terms: conditions — Neuroma, Acoustic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The surgery of a vestibular schwannoma induces balance disorders which have a an impact on the patient's daily life and disrupt their quality of life.

But the balance disorders don't seem to be the only ones factors that impaired the patient's quality of life. It has been alrealdy shown that emotional and psychological factors are also related to patient's quality of life.

This study evaluates the relationship between the balance control compensation and these factors (i.e. emotional and psychological) in the vestibular schwannoma resection process.

DETAILED DESCRIPTION:
The research protocol is based on 5 evaluation: 3 days before surgery, 8 days, 30 days, 90 days and 360 days after surgery including posturographic tests, videonystagmography and psychological questionnaires at each evaluation.

ELIGIBILITY:
Inclusion Criteria:

* patients with unilateral vestibular schwannoma (stage I to IV according to the Koos classification) with an indication for surgery.
* age between 18 and 75 years
* patients with written informed consent
* patients with Social Security affiliation

Exclusion Criteria:

* patients with psychiatrics pathologies
* ear pathology different from vestibular schwannoma (cholesteatoma of the middle ear, tympanic membrane perforation)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with vestibular schwanomma with an indication for surgery.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-08; Primary Completion 2015-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
psycholgical factors measures | one year
  The same evaluation protocole will be performed 5 times (3 days before surgery, 8 days, 30 days, 90 days and one year after surgery), with this measures:
  -score of psychological questionnaires:Revised NEO Personality Inventory (NEO PI-R), Bref Cope (coping questionnaire), Revised Illness Perception Questionnaire (IPQ-R),World Health Organisation quality of life(WHOQOL-Bref) and Hospital Anxiety and Depression Scale (HADS)
balance control performance | one year
  The same evaluation protocole will be performed 5 times (3 days before surgery, 8 days, 30 days, 90 days and one year after surgery), with the measures of the score of balance performance with sensory organisation test
vestibular performance | one year
  The same evaluation protocole will be performed 5 times (3 days before surgery, 8 days, 30 days, 90 days and one year after surgery), with the measures of the score of vestibular performance with videonystagmography

CONTACTS AND LOCATIONS:
Overall Officials: Cécile PARIETTI-WINKLER, MD, PhD, Principal Investigator — Central Hospital, Nancy, France
Locations (1):
- Centre Hospitalier Universitaire de Nancy, Nancy, Nancy, France